CLINICAL TRIAL: NCT07007195
Title: An Innovative Digitally-Delivered Olfactory Method for Reducing Cigarette Cravings and Supporting Smoking Cessation
Brief Title: Smart Olfaction App to Reduce Relapse
Acronym: SOARR
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: University of Pittsburgh (Other); University of Oklahoma (Other); Brown University (Other)
Responsible Party: Principal Investigator, Lorra Garey, Research Assistant Professor, University of Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004387
Record Dates: First submitted 2025-05-07; First posted 2025-06-05 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Nicotine Dependence
Keywords: Substance-Related Disorders; Smoking Cessation; Smartphone-Based Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: Cross-over assignment (Phase I) and Parallel assignment (Phase II)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I: Ad Libitum followed by Instructed Use of the Inspire Device (Experimental)
  Interventions: Device: Ad Libitum Use followed by Instructed Use of the Inspire Device; Drug: Nicotine replacement therapy (NRT); Device: Inspire Device
- Phase I: Instructed Use followed by Ad Libitum Use of the Inspire Device (Experimental)
  Interventions: Device: Instructed Use followed by Ad Libitum Use of the Inspire Device; Drug: Nicotine replacement therapy (NRT); Device: Inspire Device
- Phase II: Smart-T app + NRT + Inspire (Experimental)
  Interventions: Device: Smart-T Smoking Cessation App with the Inspire Device Condition; Drug: Nicotine replacement therapy (NRT); Device: Inspire Device
- Phase II: Smart-T + NRT (Active Comparator)
  Interventions: Device: Smart-T Smoking Cessation App Without the Inspire Device Condition; Drug: Nicotine replacement therapy (NRT)

INTERVENTIONS:
Device: Ad Libitum Use followed by Instructed Use of the Inspire Device — Participants in this condition will use the novel olfactory stimulation delivery system (Inspire), to smell a specific order designed to assist with smoking cessation for 7 days. Participants will then be instructed to record every urge to smoke and report times when they think they might smoke in the smartphone-based smoking cessation app, Insight™. When urges above 0 are reported, the app will instruct participants to use the Inspire device. On day 8, participants will receive a notification on the smartphone-based smoking cessation app, Insight™, to switch to the Instructed Use condition. Participants will then be instructed to use the Inspire device only when participants report a cigarette craving about 0 at each of the surveys prompted from the smartphone-based smoking cessation app, Insight™.
  Arms: Phase I: Ad Libitum followed by Instructed Use of the Inspire Device
Device: Instructed Use followed by Ad Libitum Use of the Inspire Device — Participants in this condition will use the novel olfactory stimulation delivery system (Inspire), to smell a specific order designed to assist with smoking cessation for 7 days. Participants will be instructed to use the Inspire device only when participants report a cigarette craving about 0 at each of the surveys prompted from the smartphone-based smoking cessation app, Insight™. On day 8, participants will receive a notification on the smartphone-based smoking cessation app, Insight™, to switch to the Ad Libitum condition. Participants will then control how often they use Inspire and will be instructed to record every urge to smoke and report times when they think they might smoke in the smartphone-based smoking cessation app, Insight™.
  Arms: Phase I: Instructed Use followed by Ad Libitum Use of the Inspire Device
Device: Smart-T Smoking Cessation App with the Inspire Device Condition — Smart-T provides content during the pre-quit and post-quit periods to prepare and support participants during their quit attempts. Smart-T app contains multiple components, including an EMA delivery and data transfer system, automated messages based on EMA responses, and on-demand content. Participants will use Smart-T for 13 weeks. Participants will also use the Inspire device.
  Arms: Phase II: Smart-T app + NRT + Inspire
Device: Smart-T Smoking Cessation App Without the Inspire Device Condition — Smart-T provides content during the pre-quit and post-quit periods to prepare and support participants during their quit attempts. Smart-T app contains multiple components, including an EMA delivery and data transfer system, automated messages based on EMA responses, and on-demand content. Participants will use Smart-T for 13 weeks.
  Arms: Phase II: Smart-T + NRT
Drug: Nicotine replacement therapy (NRT) — NRT patches will be provided to assist with cravings and withdrawal symptoms following the quit attempts.
Device: Inspire Device — The Inspire Device is a novel olfactory stimulation delivery system. It is a self-contained system with seven sealed chambers, with six gel matrix's that contain a distinct odor and one odorless gel matrix. Participants will press a button on the device to release an odor for participants to smell.
  Arms: Phase I: Ad Libitum followed by Instructed Use of the Inspire Device; Phase I: Instructed Use followed by Ad Libitum Use of the Inspire Device; Phase II: Smart-T app + NRT + Inspire

SUMMARY:
The proposed project aims to refine and test a novel biobehavioral smoking cessation intervention that integrates the strategic application of olfactory stimulation to reduce cigarette craving with an established smartphone-based smoking cessation application. The specific aims of this study are: (1) refine the design and methodology of our olfactory stimulation delivery system (OSDS) and (2) compare, in a pilot randomized controlled trial (RCT), the effects of a smartphone based app for smoking cessation (Smart-T) with and without the OSDS on smoking cessation outcomes.

DETAILED DESCRIPTION:
The objective of the current trial is to refine a novel biobehavioral smoking cessation intervention that integrates the strategic application of olfactory stimulation to reduce cigarette cravings (olfactory stimulation delivery system; OSDS) and then to test the OSDS as an adjunctive support for smoking cessation when integrated with an established smartphone-based smoking cessation application (Smart-T).

The study will be conducted in two phases. Phase I will consist of a crossover, micro-randomized controlled trial to inform methodology for odor administration and examine the effects of OSDS on craving reduction. Treatment-seeking smokers (N=32) will engage in a self-guided quit attempt and use the OSDS for 14 days. Using a crossover randomization design, participants will complete 7 days of ad libitum OSDS use and 7 days of instructed OSDS use. Participants will complete an initial online pre-screener, an enrollment call, a baseline survey via the app, a randomization call, and 5 daily EMAs during the study. At the end of Phase I, participants will complete a qualitative interview over Zoom and a quantitative survey in the app to assess their experiences. Phase II will be a RCT in which participants (N=100) will be randomized to either (1) Smart-T with a nicotine patch (Smart-T) or (2) Smart-T with a nicotine patch and OSDS as an adjunctive feature (Smart-T+O). Participants will complete a baseline assessment, daily EMAs for 13 weeks (1-week pre-quit and 12 weeks post-quit), a follow-up assessment at 12 weeks post-quit via the app, and a qualitative interview over Zoom. All participants will have access to Smart-T intervention materials for smoking cessation. Smoking status will be biochemically verified at multiple time points using a Carbon Monoxide monitor, which will be mailed to participants along with usage instructions.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to read, understand and speak English
* Currently smoke at least 5 cigarettes daily for one year or longer
* Do not currently smoke marijuana or currently smoke marijuana but willing to not smoke during the duration of the study
* Have an active smartphone that is Apple or Android based
* Have phone service including a data plan
* Interested in downloading the study app onto their personal phone
* Motivated to quit smoking
* Willing and able to complete study procedures
* Willing to quit smoking for 14 days (Phase I) or willing to quit smoking for 13 weeks (Phase II)

Exclusion Criteria:

* Olfactory dysfunction including inability to smell, a very weak or distorted sense of smell, or sensitivity to odors
* Report any allergies or negative reactions to odors/fragranced products
* Not being fluent in English
* Being pregnant by self-report
* Report hypertension that is not under control
* Have had a heart attack within the past two weeks
* Those who participated in Phase I will not be eligible to participate in Phase II
* Have a smartphone that is not compatible with the Insight mHealth platform
* Report using electronic cigarette or vaping device in the past 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-10-17 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
OSDS Use | Phase I: Post randomization to End of Study (14 days post-quit date)
  Descriptive data regarding use times and frequency will be assessed.
Odor Assessment | Phase I: Post randomization to End of Study (14 days post-quit date)
  Reports of odor assessment will be used to determine if sniffing specific odors reduce craving more than an odor blank.
Craving Reduction | Phase I: Post randomization to End of Study (14 days post-quit date). Phase II: Post randomization to End of Study (12 weeks post-quit date)
  Participants will report craving levels multiple times per day via the app. Reduction in craving levels over time will be analyzed.
Device Acceptability | Phase I: End of Study (14 days post-quit date). Phase II: End of Study (12 weeks post-quit date)
  Participant satisfaction ratings and qualitative feedback. Acceptability will be assessed through post-intervention surveys and qualitative interviews, focusing on perceived usefulness, ease of use, and overall satisfaction.
Smoking Abstinence | Phase II: Randomization to End of Study
  Biochemically confirmed 7-day point prevalence abstinence 12 weeks following the scheduled quit day.

CONTACTS AND LOCATIONS:
Overall Officials: Lorra Garey, Ph.D., Principal Investigator — University of Houston; Michael Businelle, Ph.D., Principal Investigator — University of Oklahoma Health Sciences; Michael Sayette, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- RESTORE Laboratory: Research on Emotion, Substance Use Treatment Outcomes, Rehabilitation, and Empowerment, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No